CLINICAL TRIAL: NCT05907200
Title: Ultrasound in Combination With Manual Therapy in the Treatment of Ischemic Digital Ulcers in Systemic Sclerosis
Brief Title: Ultrasound Therapy and Manual Therapy in Digital Ischemic Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Prof.ssa Giulia Letizia Mauro, Professor, University of Palermo
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MFR0022023
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Systemic Sclerosis
Keywords: rehabilitation; skin ulcer; ultrasound therapy; disability
MeSH Terms: conditions — Scleroderma, Systemic; Skin Ulcer | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Group (Experimental): It received rehabilitation treatment consisting of a combination of manual therapy (McMennel joint manipulation, pumping and connective tissue massage) and US water immersion.
  Interventions: Other: combination ultrasound therapy and manual therapy
- Control Group (Placebo Comparator): It received rehabilitation treatment consisting of manual therapy alone
  Interventions: Other: manual therapy

INTERVENTIONS:
Other: combination ultrasound therapy and manual therapy — The proposed manual therapy lasted 90 minutes and involved a combination of three different techniques: McMennel manipulation, connective tissue massage and mobilization technique of pumping. Patients in the treatment group also received a treatment with US (I-Tech medical device certified UT2 CE0476) in combination with manual therapy. Dipping technique was applied with a frequency of 1 MHz, intensity of 1W/cm2, duty cycle of 60% and a duration of 15 minutes per session.
  Arms: Treatment Group
Other: manual therapy — manual treatment lasting 90 minutes which involved a combination of three different techniques: McMennel manipulation, connective tissue massage and pumping mobilization technique.
  Arms: Control Group

SUMMARY:
The objective of this before-after non-randomized trial study is to evaluate the efficacy of ultrasound therapy in combination with manual therapy in the management of systemic sclerosis patients with IDU. The main questions it intends to answer are:

• Is this combination of treatments effective in these patients in terms of improvement in hand functional ability, pain relief, injury healing, and quality of life?

Participants will receive rehabilitation treatment consisting of a combination of manual therapy (McMennel joint manipulation, pumping, and connective tissue massage) and US water immersion. The researchers will compare the group of participants, called the treatment group, with a control group to see if:

• Is the combined treatment of ultrasound therapy and manual therapy more effective in these patients than manual therapy alone?

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of SSc according to the ACR and EULAR criteria
* presence of IDU in active phase
* naïve to rehabilitation treatment for their hands and upper limbs
* written in-formed consent to participate in the study.

Exclusion Criteria:

* presence of skin lesions due to other conditions (e.g., trauma);
* pregnancy;
* infectious diseases (e.g. HIV, HBV, HCV);
* myositis;
* arthritis;
* other rheumatological diseases and immunodepression.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
functional capacity | after 4 weeks of treatment
  Duruoz's hand index. The total score ranges from 0-90 with higher scores indicating poorer hand functioning.

SECONDARY OUTCOMES:
pain intensity | after 4 weeks of treatment
  numerical rating scale; the total score ranges from 0 to 10, with higher scores indicating more pain.
ulcer assessment | after 4 weeks of treatment
  Pressure Sore Status Tool; The score is between 13 and 65. Higher total scores indicated more severe wound status.
disease-related quality of life | after 4 weeks of treatment
  The 36-Item Short Form Health Survey; The score ranges from 0 to 100, where higher scores indicate improved health.

CONTACTS AND LOCATIONS:
Locations (1):
- Functional Recovery and Rehabilitation Unit of the A.O.U.P. Paolo Giaccone, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No